CLINICAL TRIAL: NCT01118364
Title: Effect of Cannabis on Simulated and Actual Driving in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Assistance Publique Hôpitaux de Marseille, direction de la recherche
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2009-A00940-57; 2009/24 (Registry Identifier: internal reference)
Record Dates: First submitted 2010-05-05; First posted 2010-05-06 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
Keywords: Social circumstances
MeSH Terms: interventions — nabiximols; Tobacco Products

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- cigarette with cannabis (Experimental): a cigarette tobacco trade mark "Drum" with the addition of 250 mg of cannabis resin with 8% of D9THC (20 mg per cigarette)
  Interventions: Other: Cannabis
- cigarette without cannabis (Other): a cigarette tobacco trade mark "Drum"
  Interventions: Other: tobacco

INTERVENTIONS:
Other: Cannabis — a cigarette tobacco trade mark "Drum" with the addition of 250 mg of cannabis resin with 8% of D9THC (20 mg per cigarette)45 minutes before simulating or real driving
  Arms: cigarette with cannabis
Other: tobacco — a cigarette tobacco trade mark "Drum" 45 minutes before simulating or real driving
  Arms: cigarette without cannabis

SUMMARY:
Assess the effect of cigarette smoking of tobacco with or without addition of resin cannabis on driving performance in healthy volunteers in simulated driving in Marseille and Toulouse, and in real world driving to Bordeaux.

Multicenter Study of phase 1, randomized, double-blind, cross plan, carried out in healthy male volunteers.

DETAILED DESCRIPTION:
* To compare performance data driving with the data self-assessed on the ability to drive, and the level of sleepiness and fatigue
* To measure the effects of distractive task on driving performance, consisting of a conversation with co-driver of the real or simulated vehicle (a series of difficult questions involving reflection)
* To validate the (known) effects of cannabis
* To adapt equipment and standardize methods for the pharmacological studies evaluating other types of substances having an impact on driving (antihistamines, antidepressants, antiparkinsonian ...) and other populations of subjects (men versus women, young versus elderly, healthy versus sick ...)
* To compare data obtained under conditions of simulated driving and actual driving situation, under identical experimental conditions (volunteers, narcotic substance, experimental) and measure the degree of ecological validity of the simulation of driving

ELIGIBILITY:
Inclusion Criteria:

* Weight +/- 10% of ideal weight
* Tobacco smoker moderate
* Having already smoked of the cannabis (less 1 time per month)
* Not consuming in a way exaggerated by some coffee, tea or cola
* Not having acute or chronic pathologies
* Normal electrocardiogram
* Not taking a drug interfering with the study
* Not presenting disorder of sleeping
* Having a driving license for at least 3 years and driving more 3000 km per year
* Normal acuteness or corrected visual acuteness and normal vision of colors
* Reachable and available during the study
* No nausea or vomit during using of a driving simulator
* Having a national insurance scheme
* Volunteer

Exclusion Criteria:

* Women
* Weight deviating of 10% of ideal weight
* Consuming moreover 5 cup of caffeine drinks
* Drinking alcohol regularly
* Acute or chronic pathologies interfering with the study
* Abnormal electrocardiogram
* Asthmatic
* Dependence present or spent in a psychotropic substance
* Presenting an anxious or depressive syndrome
* Circadian typology (Horne et Ostberg)
* Positive control in the cannabis in urines the day of the balance assessment of inclusion
* Positive control in alcohol the day of the balance assessment of inclusion
* Participating in another clinical study
* Having collected an upper total amount of compensations allowances
* Deprived of freedom further to a court or administrative order
* Risk of not observance
* Duration average of sleep of 3 nights previous every session lower than 80 % of the average duration of sleep which the volunteer thinks of needing to be in shape

Ages: 25 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-05; Primary Completion 2011-02 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Line crossing | 1 years
  Measurement of inappropriate crossing of the limits of track in real or simulated driving

SECONDARY OUTCOMES:
Weaving | 1 years
  Measure of the deviation of the lateral position of the vehicle on the real or simulated road
Evaluation of sleepiness and fatigue | 1 years
Evaluation of fitness to drive | 1 years
Evaluation of fitness to drive during work distraction | 1 years

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Hôpitaux de Marseille, Marseille, France